CLINICAL TRIAL: NCT03084003
Title: Effects of Almond Consumption on Cardiovascular, Metabolomic, and Microbiome Profiles in Millennials: Implications of Systemic Glucoregulatory Mechanisms
Brief Title: Effects of Almond Consumption on Cardiovascular, Metabolomic, and Microbiome Profiles in Millennials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Merced (Other)
Responsible Party: Principal Investigator, Rudy Ortiz, Professor, University of California, Merced
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UCM2016-86
Record Dates: First submitted 2017-02-21; First posted 2017-03-20 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Diet Intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Almond group (Experimental): 2 oz. of almonds everyday for 8 weeks
  Interventions: Dietary Supplement: Almonds
- Control group (Active Comparator): Isoenergetic control group 5 graham cracker sheets everyday for 8 weeks
  Interventions: Dietary Supplement: Graham crackers

INTERVENTIONS:
Dietary Supplement: Almonds
  Arms: Almond group
Dietary Supplement: Graham crackers
  Arms: Control group

SUMMARY:
The purpose of the study is to examine the effects of almond snacking on metabolic, cardiovascular and microbiome profiles in college freshmen.

DETAILED DESCRIPTION:
Nut (principally almond) consumption helps ameliorate cardiovascular disease, reduce the risk of type II diabetes mellitus (T2DM). Recent studies have demonstrated improvements in glycemic control in T2DM and impaired glucose tolerant (IGT) subjects as well as in healthy adults. The association between nut consumption and diabetes prevalence is largely mediated by changes in body mass (adiposity). The application of metabolomic and lipidomic approaches to better asses the mechanisms regulating carbohydrates and lipids in an almond-based study has not been performed.

Additionally, the gut microbiota has been proposed to contribute to a number of metabolic disorders including insulin sensitivity, glucose metabolism, and other cardiometabolic risk factors. However, data demonstrating the complex interactions among dietary interventions, gut microbiome, glucose regulation, and cardiovascular phenotype are lacking.

Furthermore, because all the studies on nut consumption and health have been performed on adults (median age of subjects: +40 years) and given the increasing incidence of metabolic disorders (obesity, insulin resistance, etc.) at much younger stages of life especially in the Central Valley of California, no data exist on the potential benefits of almonds in ameliorating metabolic disorders at a much earlier life stage. This may be clinically more important than studies in adults because the transition from adolescence to adulthood is associated with a number of potential risk factors unique to this age group, especially in those that enter their first year of college. The fixed age of the participants contributes to a more homogeneous population than has been previously studied, which greatly minimizes the potential for age-dependent alterations in physiology to either potentiate or mask the effects of the almonds on metabolic mechanisms. The nutritional independence that is associated with going away to college poses many potential health challenges, for example the phenomenon, "Freshman 15". The increased prevalence of overweight and obesity is greatest in 18-29 year olds, especially among those reporting some college education (10.6%-17.8% vs 7.1%-12.1% in 18-29 year olds overall) suggesting that some aspect of the collegiate experience is associated with weight gain.

While almond-supplemented diets have been shown to reduce body mass or ameliorate weight gain, the evidence substantiating the benefits of functional foods in addressing the weight gain commonly associated with the transition to college is scarce and an untapped area of research. Furthermore, this transition to nutritional independence makes new college students vulnerable to additional alterations in eating patterns. Among these concerns are the relatively high number of college freshmen that reported skipping breakfast (20%-43%), which is by far the most skipped meal among those studies reviewed. This is important because chronically skipping breakfast in adolescents has detrimental outcomes on cardiometabolic health and has negative impacts on academic performance. Additionally, most college students snack, with snacking common both in the morning and the afternoon. Data suggest a benefit to snacking on peanuts and almonds. However, the benefits of snacking in young college students who routinely skip a meal (breakfast here) are not defined. Therefore, being able to demonstrate the benefits of almonds in college "breakfast skippers" would have significant implications for young adults in their first year of college, and thus, provide an ideal opportunity to further address this line of inquiry. Lastly, the application of metabolomic and lipidomic approaches to better assess the mechanisms regulating carbohydrates and lipids in an almond-based study has not been performed. Advancements in high-throughput analytical techniques have initiated a renaissance in the study of metabolism on a grand scale that allow for robust assessment of nutritional status and cellular responses. These approaches provide an advantage of mapping metabolites in such a fashion that changes in mechanisms can be elucidated as demonstrated by the SuGAR Project.

ELIGIBILITY:
* Inclusion Criteria:

  * 18-22 years of age
  * Newly enrolled, 1st-year college students at University of California, Merced
  * Willing to eat almonds and study snacks
  * Willing to comply with the study protocol
  * Consistent diet and activity patterns
  * Non-smoker >1 year or more
* Exclusion Criteria:

  * Nut allergies
  * Illicit drug use
  * Medications that affect metabolism or appetite
  * Anti-inflammatory medications, analgesics and antibiotics
  * Diabetes or pre-diabetes, uncontrolled hypertension, cardiovascular disease or dyslipidemia requiring drug therapy
  * Gastrointestinal disease and/or bariatric surgery

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Change in fasting blood glucose | Change from baseline at 8 weeks
2-hour oral glucose tolerance test | At the end of 8 week intervention
Change in fasting blood insulin | Change from baseline at 8 weeks
Change in stool microbiome profiles | Change from baseline at 8 weeks

SECONDARY OUTCOMES:
Weight | Every 2 weeks over the 8 week intervention
Body composition | Every 2 weeks over the 8 week intervention
Waist circumference | Every 2 weeks over the 8 week intervention
Blood pressure | Every 2 weeks over the 8 week intervention
24-hour appetite ratings | Baseline, 4 weeks into intervention and end of 8 week intervention
Hip circumference | Every 2 weeks over the 8 week intervention
Flow Mediated Dilation (FMD) | At the end of 8 week intervention
  As a measure of endothelial function
Urinary 8-isoprostane | Baseline and end of 8 week intervention
Urinary electrolytes | Baseline and end of 8 week intervention
Urinary angiotensinogen | Baseline and end of 8 week intervention
Urinary creatinine clearance | Baseline and end of 8 week intervention
Fasting lipid profile | Baseline, 4 weeks into intervention and end of 8 week intervention
Physical activity | Baseline, 4 weeks into intervention and end of 8 week intervention
  Research Tracker 6 (RT6) accelerometers
Hepatic glucose metabolism | End of 8 week intervention
  Isotopic dilution

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Ortiz, PhD, Principal Investigator — UNIV OF CALIFORNIA MERCED
Locations (1):
- University of California, Merced, Merced, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abazarfard Z, Salehi M, Keshavarzi S. The effect of almonds on anthropometric measurements and lipid profile in overweight and obese females in a weight reduction program: A randomized controlled clinical trial. J Res Med Sci. 2014 May;19(5):457-64. PMID 25097630
- [Background] Adams SH, Hoppel CL, Lok KH, Zhao L, Wong SW, Minkler PE, Hwang DH, Newman JW, Garvey WT. Plasma acylcarnitine profiles suggest incomplete long-chain fatty acid beta-oxidation and altered tricarboxylic acid cycle activity in type 2 diabetic African-American women. J Nutr. 2009 Jun;139(6):1073-81. doi: 10.3945/jn.108.103754. Epub 2009 Apr 15. PMID 19369366
- [Background] Berkey CS, Rockett HR, Gillman MW, Field AE, Colditz GA. Longitudinal study of skipping breakfast and weight change in adolescents. Int J Obes Relat Metab Disord. 2003 Oct;27(10):1258-66. doi: 10.1038/sj.ijo.0802402. PMID 14513075
- [Background] Brevard PB, Ricketts CD. Residence of college students affects dietary intake, physical activity, and serum lipid levels. J Am Diet Assoc. 1996 Jan;96(1):35-8. doi: 10.1016/S0002-8223(96)00011-9. PMID 8537567
- [Background] Cani PD, Delzenne NM. Gut microflora as a target for energy and metabolic homeostasis. Curr Opin Clin Nutr Metab Care. 2007 Nov;10(6):729-34. doi: 10.1097/MCO.0b013e3282efdebb. PMID 18089955
- [Background] Cohen AE, Johnston CS. Almond ingestion at mealtime reduces postprandial glycemia and chronic ingestion reduces hemoglobin A(1c) in individuals with well-controlled type 2 diabetes mellitus. Metabolism. 2011 Sep;60(9):1312-7. doi: 10.1016/j.metabol.2011.01.017. Epub 2011 Apr 12. PMID 21489570
- [Background] Devitt AA, Kuevi A, Coelho SB, Lartey A, Lokko P, Costa N, Bressan J, Mattes RD. Appetitive and Dietary Effects of Consuming an Energy-Dense Food (Peanuts) with or between Meals by Snackers and Nonsnackers. J Nutr Metab. 2011;2011:928352. doi: 10.1155/2011/928352. Epub 2011 Jan 22. PMID 21808728
- [Background] Diamant M, Blaak EE, de Vos WM. Do nutrient-gut-microbiota interactions play a role in human obesity, insulin resistance and type 2 diabetes? Obes Rev. 2011 Apr;12(4):272-81. doi: 10.1111/j.1467-789X.2010.00797.x. Epub 2010 Aug 26. PMID 20804522
- [Background] Driskell JA, Kim YN, Goebel KJ. Few differences found in the typical eating and physical activity habits of lower-level and upper-level university students. J Am Diet Assoc. 2005 May;105(5):798-801. doi: 10.1016/j.jada.2005.02.004. PMID 15883559
- [Background] Fiehn O, Garvey WT, Newman JW, Lok KH, Hoppel CL, Adams SH. Plasma metabolomic profiles reflective of glucose homeostasis in non-diabetic and type 2 diabetic obese African-American women. PLoS One. 2010 Dec 10;5(12):e15234. doi: 10.1371/journal.pone.0015234. PMID 21170321
- [Background] Grapov D, Adams SH, Pedersen TL, Garvey WT, Newman JW. Type 2 diabetes associated changes in the plasma non-esterified fatty acids, oxylipins and endocannabinoids. PLoS One. 2012;7(11):e48852. doi: 10.1371/journal.pone.0048852. Epub 2012 Nov 8. PMID 23144998
- [Background] Heatherton TF, Nichols P, Mahamedi F, Keel P. Body weight, dieting, and eating disorder symptoms among college students, 1982 to 1992. Am J Psychiatry. 1995 Nov;152(11):1623-9. doi: 10.1176/ajp.152.11.1623. PMID 7485625
- [Background] Hoffman DJ, Policastro P, Quick V, Lee SK. Changes in body weight and fat mass of men and women in the first year of college: A study of the "freshman 15". J Am Coll Health. 2006 Jul-Aug;55(1):41-5. doi: 10.3200/JACH.55.1.41-46. PMID 16889314
- [Background] Josse AR, Kendall CW, Augustin LS, Ellis PR, Jenkins DJ. Almonds and postprandial glycemia--a dose-response study. Metabolism. 2007 Mar;56(3):400-4. doi: 10.1016/j.metabol.2006.10.024. PMID 17292730
- [Background] Li SC, Liu YH, Liu JF, Chang WH, Chen CM, Chen CY. Almond consumption improved glycemic control and lipid profiles in patients with type 2 diabetes mellitus. Metabolism. 2011 Apr;60(4):474-9. doi: 10.1016/j.metabol.2010.04.009. Epub 2010 May 23. PMID 20580779
- [Background] Luo C, Zhang Y, Ding Y, Shan Z, Chen S, Yu M, Hu FB, Liu L. Nut consumption and risk of type 2 diabetes, cardiovascular disease, and all-cause mortality: a systematic review and meta-analysis. Am J Clin Nutr. 2014 Jul;100(1):256-69. doi: 10.3945/ajcn.113.076109. Epub 2014 May 21. PMID 24847854
- [Background] Mokdad AH, Serdula MK, Dietz WH, Bowman BA, Marks JS, Koplan JP. The spread of the obesity epidemic in the United States, 1991-1998. JAMA. 1999 Oct 27;282(16):1519-22. doi: 10.1001/jama.282.16.1519. PMID 10546690
- [Background] Mori AM, Considine RV, Mattes RD. Acute and second-meal effects of almond form in impaired glucose tolerant adults: a randomized crossover trial. Nutr Metab (Lond). 2011 Jan 28;8(1):6. doi: 10.1186/1743-7075-8-6. PMID 21276226
- [Background] Quehenberger O, Armando AM, Brown AH, Milne SB, Myers DS, Merrill AH, Bandyopadhyay S, Jones KN, Kelly S, Shaner RL, Sullards CM, Wang E, Murphy RC, Barkley RM, Leiker TJ, Raetz CR, Guan Z, Laird GM, Six DA, Russell DW, McDonald JG, Subramaniam S, Fahy E, Dennis EA. Lipidomics reveals a remarkable diversity of lipids in human plasma. J Lipid Res. 2010 Nov;51(11):3299-305. doi: 10.1194/jlr.M009449. Epub 2010 Jul 29. PMID 20671299
- [Background] Rodriguez R, Mowrer J, Romo J, Aleman A, Weffer SE, Ortiz RM. Ethnic and gender disparities in adolescent obesity and elevated systolic blood pressure in a rural US population. Clin Pediatr (Phila). 2010 Sep;49(9):876-84. doi: 10.1177/0009922810368135. Epub 2010 Jun 3. PMID 20522603
- [Background] Smith KJ, Gall SL, McNaughton SA, Blizzard L, Dwyer T, Venn AJ. Skipping breakfast: longitudinal associations with cardiometabolic risk factors in the Childhood Determinants of Adult Health Study. Am J Clin Nutr. 2010 Dec;92(6):1316-25. doi: 10.3945/ajcn.2010.30101. Epub 2010 Oct 6. PMID 20926520
- [Background] Tan SY, Mattes RD. Appetitive, dietary and health effects of almonds consumed with meals or as snacks: a randomized, controlled trial. Eur J Clin Nutr. 2013 Nov;67(11):1205-14. doi: 10.1038/ejcn.2013.184. Epub 2013 Oct 2. PMID 24084509
- [Background] Vella-Zarb RA, Elgar FJ. The 'freshman 5': a meta-analysis of weight gain in the freshman year of college. J Am Coll Health. 2009 Sep-Oct;58(2):161-6. doi: 10.1080/07448480903221392. PMID 19892653
- [Background] Wien MA, Sabate JM, Ikle DN, Cole SE, Kandeel FR. Almonds vs complex carbohydrates in a weight reduction program. Int J Obes Relat Metab Disord. 2003 Nov;27(11):1365-72. doi: 10.1038/sj.ijo.0802411. PMID 14574348
- [Background] Zivkovic AM, German JB. Metabolomics for assessment of nutritional status. Curr Opin Clin Nutr Metab Care. 2009 Sep;12(5):501-7. doi: 10.1097/MCO.0b013e32832f1916. PMID 19584717
- [Derived] Dhillon J, Pandey S, Newman JW, Fiehn O, Ortiz RM. Almond consumption for 8 weeks differentially modulates metabolomic responses to an acute glucose challenge compared to crackers in young adults. Nutr Res. 2025 Mar;135:67-81. doi: 10.1016/j.nutres.2025.01.003. Epub 2025 Jan 8. PMID 39965269
- [Derived] Dhillon J, Pandey S, Newman JW, Fiehn O, Ortiz RM. Metabolic Responses to an Acute Glucose Challenge: The Differential Effects of Eight Weeks of Almond vs. Cracker Consumption in Young Adults. medRxiv [Preprint]. 2024 May 20:2024.05.19.24307571. doi: 10.1101/2024.05.19.24307571. PMID 38826341
- [Derived] Dhillon J, Newman JW, Fiehn O, Ortiz RM. Almond Consumption for 8 Weeks Altered Host and Microbial Metabolism in Comparison to a Control Snack in Young Adults. J Am Nutr Assoc. 2023 Mar-Apr;42(3):242-254. doi: 10.1080/07315724.2021.2025168. Epub 2022 Feb 23. PMID 35512761
- [Derived] Dhillon J, Li Z, Ortiz RM. Almond Snacking for 8 wk Increases Alpha-Diversity of the Gastrointestinal Microbiome and Decreases Bacteroides fragilis Abundance Compared with an Isocaloric Snack in College Freshmen. Curr Dev Nutr. 2019 Jul 3;3(8):nzz079. doi: 10.1093/cdn/nzz079. eCollection 2019 Aug. PMID 31528836
- See also: Nuts for diabetes prevention and management — http://www.fda.gov.tw/upload/189/Content/2014012817285169148.pdf
- See also: Adolescent Health in the United States, 2007 — https://www.cdc.gov/nchs/data/misc/adolescent2007.pdf
- See also: Reduced physical activity levels associated with obesity in rural Hispanic adolescent females. — http://online.liebertpub.com/doi/abs/10.1089/chi.2011.0007